CLINICAL TRIAL: NCT04804098
Title: The Effect of Rate (Slope) of Compression on the Incidence of Symptomatic Eustachian Tube Dysfunction and Middle Ear Barotrauma: a Phase III Prospective Study.
Brief Title: Effect of Rate (Slope) of Compression on the Incidence of Symptomatic ETD and MEB: a Phase III Prospective Study.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Owen J O'Neill, MD, MPH, Medical Director Division of Undersea & Hyperbaric Medicine, Northwell Health
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Compression Hyperbaric III
Record Dates: First submitted 2021-02-10; First posted 2021-03-18 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Ear Barotrauma; Middle Ear Disease; Ear Diseases; Pressure Injury; Eustachian Tube Dysfunction; Middle Ear; Injury; Middle Ear Barotrauma
Keywords: Ear Pressure; Otic Barotrauma; Hyperbaric; Pressure Equalization; O'Neill Grading System; Compression Rate
MeSH Terms: conditions — Ear Diseases; Pressure Ulcer; Wounds and Injuries | interventions — Appointments and Schedules

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 15 Minute Non-linear Compression Profile (Active Comparator): Compression Profile/Schedule 1 = 15 minute non-linear, Total Time Interval of Compression to treatment depth = 15 minutes Rate (slope) of compression = Non-Linear rate of compression = 2 fsw/min to a depth of 13 fsw, then 3 fsw/min up to a depth of 35 fsw, then 5 fsw/min to arrival at the treatment depth of 45 fsw
  Interventions: Procedure: Compression Profile/Schedule: 15 minute Non-Linear compression from start of the daily treatment until treatment pressure is reached (45 fsw)
- 15 Minute Linear Compression Profile (Active Comparator): Compression Profile/Schedule 2 = 15 minute linear, Total Time Interval of Compression to treatment depth = 15 minutes Rate (slope) of compression = Linear rate of compression = 4.5 fsw/min to arrival at the treatment depth 45 fsw
  Interventions: Procedure: Compression Profile/Schedule: 15 minute Linear compression from start of the daily treatment until treatment pressure is reached (45 fsw)

INTERVENTIONS:
Procedure: Compression Profile/Schedule: 15 minute Non-Linear compression from start of the daily treatment until treatment pressure is reached (45 fsw) — Patients will be compressed according to the 15 minute non-linear compression schedule on a rotating daily basis. A total of 2 randomized hyperbaric treatment compression profiles (accepted standards of care) will be alternated over the patients course of treatment on a daily basis daily to the prescribed treatment depth. There are multiple patients exposed during the compression profile randomized for that day. The patients are exposed over the course of 4-12 weeks using one of the two compression protocols to be studied on alternating days.
  Other Names: Hyperbaric Compression Schedule 15 min non-linear
  Arms: 15 Minute Non-linear Compression Profile
Procedure: Compression Profile/Schedule: 15 minute Linear compression from start of the daily treatment until treatment pressure is reached (45 fsw) — Patients will be compressed according to the 15 minute linear compression schedule on a rotating daily basis with compression. A total of 2 randomized hyperbaric treatment compression profiles (accepted standards of care) will be alternated over the patients course of treatment on a daily basis daily to the prescribed treatment depth. There are multiple patients exposed during the compression profile randomized for that day. The patients are exposed over the course of 4-12 weeks using one of the two compression protocols to be studied on alternating days.
  Other Names: Hyperbaric Compression Schedule 15 min linear
  Arms: 15 Minute Linear Compression Profile

SUMMARY:
Eustachian tube dysfunction (ETD) and middle ear barotrauma (MEB) are common reported complications during hyperbaric oxygen treatment. The Phase I study data was the first to demonstrate a statistically significant decrease in the occurrence of symptomatic ETD and middle ear barotrauma (MEB). The Phase I Trial suggested the total time interval and rate (slope) of compression (ROC) may be a determining factor in ETD and MEB. This Phase II study investigates an optimal total time interval and rate of compression to reduce ETD and MEB when considering each multiplace treatment (with multiple patients) as the unit of observation collectively as a group, rather than for each individual patient.

Data will be collected prospectively on group patient-treatment exposures. Our investigators randomly assign patient-treatment group exposures to two different rates (slopes) of compression. These are limited to the linear versus the non-linear rates (slopes) of compression identical to two of four compression profiles used in the Phase I and Phase II trials. All patients experiencing symptoms of ETD and MEB requiring compression stops will be evaluated post treatment to confirm the presence of ETD and MEB using the O'Neill Grading System (OGS). Data will be analyzed using the IBM-SPSS statistical software program.

The number of compression holds observed in each of the compression schedules/compression profiles using an identical 15-minute total time interval of compression but varying in the rate (slope) of compression will be recorded as in the Phase I and II studies. Symptomatic patients who required compression stops (as in the Phase I trial) using a USN TT 9 during elective hyperbaric oxygen treatments in a Class A multiplace hyperbaric chamber will be compared. Statistical analysis using descriptive and Inferential statistics will be applied to the patients requiring first stops in the compression profiles. This will be used to further evaluate the data restricted to the rate of compression (linear vs. non-linear) and whether this is associated with the number of compression holds. The 15-minute total time interval of compression will be identical in both compression profiles studied since this was found to be the total time interval of compression with the least number of treatment stops/holds in the phase I and phase II studies.

DETAILED DESCRIPTION:
Eustachian tube dysfunction (ETD) and middle ear barotrauma (MEB) are common reported complications during hyperbaric oxygen treatment. The Phase I study data was the first to demonstrate a statistically significant decrease in the occurrence of symptomatic ETD and middle ear barotrauma (MEB) in specific compression profiles among those used as common standards of care in hyperbaric oxygen treatment. The Phase I Trial suggested the total time interval and rate (slope) of compression (ROC) may be a determining factor in ETD and MEB. The Phase II study investigated tested the robustness of these findings with a larger sample size and failed to determine an optimal rate of compression to reduce ETD and MEB when considering each multiplace treatment (with multiple patients) as the unit of observation collectively as a group, rather than for each individual patient. In this phase III trial we will increase sample size further to determine if the effect size of the rate (slope) of compression is smaller than anticipated in the phase I and II studies requiring a larger sample size and greater power. This study will be restricted to the two compression profiles limited to the 15 minute total time interval of compression which was found to be the time interval associated with the least number of treatment holds or stops.

Data will be collected prospectively on group patient-treatment exposures. The investigators will randomly assign patient-treatment group exposures to a single identical time interval but different rates (slopes) of compression. These compression rates (slopes) were identical to those used in the Phase I and II trials. All patients experiencing symptoms of ETD and MEB requiring compression stops or holds will be evaluated post-treatment to confirm the presence of ETD and MEB using the O'Neill Grading System (OGS) for ETD/MEB.

For approximately 10 years, the investigators hyperbaric center used a routine daily multiplace chamber treatment protocol to a depth of 45 feet of seawater (fsw) (modified U.S. Navy Treatment Table 9). The chamber was compressed over a 10-minute time interval representing a 4.5 fsw/minute uniform rate of compression. This 4.5-fsw/minute compression rate throughout the total 10-minute time interval of treatment was used as a baseline compression rate to compare all other compression schedules [total compression time interval/compression rates (slopes)]. The investigators will prospectively collect data on patient-treatment group exposures after formalizing two different compression schedules each including a unique compression rate (slope) linear vs. non-linear but using the same 15-minute time interval of compression. This was similar to the Phase I and Phase II study but limited to two compression profiles.

Data will be collected prospectively on all patients receiving treatment from September 1, 2021, and October 31, 2023, and combined with the data obtained in the Phase I and II trials collected from September 8, 2014 to September 8, 2016; and February 11, 2019, and February 10, 2020 respectively. This Phase III study defines the unit of observations as a multiplace patient-treatment group exposure rather than individual patient treatment exposures. This approach was considered appropriate as a treatment stop or hold in a multiplace chamber affects all other patient occupants in the same treatment group exposure. It results in a hold for all patients in the multiplace chamber during that respective treatment. The possible effects on the other patients in the same treatment group could possibly confound our outcomes. The effect of rate (slope) of compression on an individual patient can be better ascertained at the individual patient level in a monoplace chamber, without influencing the effect on other patients.

To mitigate the risk of confounding, only the first stop will be used as the stop or hold indicator for that particular patient-treatment group exposure. Data will be collected on the patient(s) experiencing the stop or hold. All patients will undergo pre-treatment video otoscopy with baseline tympanic membrane (TM) photos and video of TM motion documenting the patients ability to equalize. This is used to assess potential Eustachian tube patency and proper equalization performance to help exclude individual patient technique as a confounding variable. Photos will be repeated at the end of treatment on any patient(s) complaining of symptoms referable to ETD/MEB that require a stop during compression.

Multiple stops for the same patient on the same treatment will not be considered. Only the first compression stop or hold during each treatment exposure will be recorded or assigned as a patient-treatment stop representing that particular patient-treatment group exposure. Compression stops will be made when any patient experiences difficulty equalizing (requests a stop or complains of ear discomfort of any type).

Repeat video otoscopy will be conducted on all patients complaining of symptoms referable to ETD or MEB to objectively document the grade of barotrauma at the end of the treatment. The O'Neill Grading System will be used to record the severity of the ETD or MEB. The depth of the stop, the treatment number for that particular patient, and the actions taken to alleviate the symptoms during equalization will be recorded.

The depth of the compression stop will be recorded in feet of seawater (fsw) as will be the ascent (fsw) required for the patient to clear the middle ear pressure and relieve the symptoms. The patients symptoms must be resolved, rendering the patient asymptomatic and able to continue the treatment compression profile. All team members (physicians, nurses, and technicians) present and working on the day of the exposure, are responsible for viewing the patients pre and post tympanic membrane photos and determining the grade of barotrauma using the OGS criteria.

All stops were categorized under the respective compression protocol used for that particular patient-treatment group exposure. Data will then compared using both descriptive and inferential statistical analysis including the risk difference, odds ratio (OR), two-tailed Chi Square analysis using α=0.05, and outcomes will be studied separately in a logistic regression analysis.

ELIGIBILITY:
Inclusion Criteria:

- Any patient meeting the proper diagnosis and indications to be treated with hyperbaric oxygen.

Exclusion Criteria:

* Any patient with absolute contraindications to hyperbaric oxygen treatment
* Patients with chronic bilateral perforation of the tympanic membrane or;
* A history of prior surgical placement of myringotomy tubes.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Hyperbaric oxygen chamber Treatment Stops/Holds during compression | Patients are assessed during each hyperbaric chamber compression until reaching treatment pressure/depth daily throughout the entire treatment course that varies based on diagnosis over 4-12 weeks
  Hyperbaric oxygen treatment (HBOT) protocols include a compression phase. Pressure is increased until final treatment pressure is achieved. Pressure changes vary between 14.7 psi to 35 psi. Patients experience symptoms of pain or pressure in the middle ear space because they cannot clear middle ear pressure upon compression of the chamber. Pressure symptoms are time related but not as yet slope related. Using varying rates of pressure may decrease discomfort related to clearing middle ear pressure known as Eustachian tube dysfunction (ETD) and middle ear barotrauma (MEB). They are the most common adverse effects of HBOT. The authors believe a change in slope rate of compression may decrease the occurrence of stops and decrease the incidence of ETD and MEB during HBOT. Decreasing rate of compression may further mitigate risk and decrease the incidence of symptomatic ETD and MEB.
Severity of ETD/MEB when a patient has a stop/hold during compression | Patients are assessed during each hyperbaric chamber compression until reaching treatment pressure/depth daily throughout the entire treatment course that varies based on diagnosis over 4-12 weeks
  Photo otoscopy and the severity of eustachian tub dysfunction and/or middle ear barotrauma will be defined using the O'Neill Grading System when a patient experiences a stop or hold during the compression phase of hyperbaric oxygen treatment.
  O'Neill Grading System:
  0 = Symptoms of Eustachian tube dysfunction with no objective signs of barotrauma on otoscopy
  1. = Objective evidence indicating the presence of erythema, air trapping or serous/serosanguinous effusion
  2. = Any frank bleeding in the middle ear space, tympanic membrane, external ear canal, or perforation

CONTACTS AND LOCATIONS:
Overall Officials: Owen J O'Neill, MD, MPH, Principal Investigator — Phelps Hospital Northwell Health; David Dayya, DO, PhD, MPH, Principal Investigator — Phelps Hospital Northwell Health
Locations (1):
- Phelps Hospital Northwell Health, Sleepy Hollow, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Would consider if other researchers are studying similar research question and interested in collaboration.
Supporting Information: Study Protocol, CSR
Time Frame: Post publication
Access Criteria: Contact Primary Investgators by Email

REFERENCES:
- [Background] Beuerlein M, Nelson RN, Welling DB. Inner and middle ear hyperbaric oxygen-induced barotrauma. Laryngoscope. 1997 Oct;107(10):1350-6. doi: 10.1097/00005537-199710000-00011. PMID 9331312
- [Background] Camporesi EM. Side effects of hyperbaric oxygen therapy. Undersea Hyperb Med. 2014 May-Jun;41(3):253-7. PMID 24984321
- [Background] Heyboer M 3rd, Wojcik SM, Grant WD, Chambers P, Jennings S, Adcock P. Middle ear barotrauma in hyperbaric oxygen therapy. Undersea Hyperb Med. 2014 Sep-Oct;41(5):393-7. PMID 25558548
- [Background] Lima MA, Farage L, Cury MC, Bahamad F Junior. Update on middle ear barotrauma after hyperbaric oxygen therapy-insights on pathophysiology. Int Arch Otorhinolaryngol. 2014 Apr;18(2):204-9. doi: 10.1055/s-0034-1366974. Epub 2014 Feb 10. PMID 25992091
- [Background] Ng AWA, Muller R, Orton J. Incidence of middle ear barotrauma in staged versus linear chamber compression during hyperbaric oxygen therapy: a double blinded, randomized controlled trial. Undersea Hyperb Med. 2017 Mar-Apr;44(2):101-107. doi: 10.22462/3.4.2017.3. PMID 28777900
- [Background] Plafki C, Peters P, Almeling M, Welslau W, Busch R. Complications and side effects of hyperbaric oxygen therapy. Aviat Space Environ Med. 2000 Feb;71(2):119-24. PMID 10685584
- [Background] Toklu AS, Shupak A, Yildiz S, Aktas S, Ertracht O, Ay H, Adir Y, Cimsit M. Aural barotrauma in submarine escape: is mastoid pneumatization of significance? Laryngoscope. 2005 Jul;115(7):1305-9. doi: 10.1097/01.MLG.0000165804.09586.B6. PMID 15995526
- [Background] Vahidova D, Sen P, Papesch M, Zein-Sanchez MP, Mueller PH. Does the slow compression technique of hyperbaric oxygen therapy decrease the incidence of middle-ear barotrauma? J Laryngol Otol. 2006 Jun;120(6):446-9. doi: 10.1017/S002221510600079X. PMID 16772053
- [Background] Varughese L, O'Neill OJ, Marker J, Smykowski E, Dayya D. The effect of compression rate and slope on the incidence of symptomatic Eustachian tube dysfunction leading to middle ear barotrauma: a Phase I prospective study. Undersea Hyperb Med. 2019 Mar-Apr-May;46(2):95-100. PMID 31051053
- [Background] Bove AA. Diving medicine. Am J Respir Crit Care Med. 2014 Jun 15;189(12):1479-86. doi: 10.1164/rccm.201309-1662CI. PMID 24869752
- [Background] Fitzpatrick DT, Franck BA, Mason KT, Shannon SG. Risk factors for symptomatic otic and sinus barotrauma in a multiplace hyperbaric chamber. Undersea Hyperb Med. 1999 Winter;26(4):243-7. PMID 10642071
- [Background] Goplen FK, Gronning M, Aasen T, Nordahl SH. Vestibular effects of diving - a 6-year prospective study. Occup Med (Lond). 2010 Jan;60(1):43-8. doi: 10.1093/occmed/kqp148. Epub 2009 Oct 23. PMID 19854795
- [Background] Hadanny A, Meir O, Bechor Y, Fishlev G, Bergan J, Efrati S. Seizures during hyperbaric oxygen therapy: retrospective analysis of 62,614 treatment sessions. Undersea Hyperb Med. 2016 Jan-Feb;43(1):21-8. PMID 27000010
- [Background] Mozdzanowski C, Perdrizet GA. Peripheral neuropathy may increase the risk for asymptomatic otic barotrauma during hyperbaric oxygen therapy: research report. Undersea Hyperb Med. 2014 Jul-Aug;41(4):267-72. PMID 25109078
- [Background] Sanders RW. Controlling the rate of middle ear barotrauma: an editorial perspective. Undersea Hyperb Med. 2014 Sep-Oct;41(5):355-6. No abstract available. PMID 25558542
- [Background] O'Neill OJ, Weitzner ED. The O'Neill grading system for evaluation of the tympanic membrane: A practical approach for clinical hyperbaric patients. Undersea Hyperb Med. 2015 May-Jun;42(3):265-71. PMID 26152108
- [Background] Nasole E, Zanon V, Marcolin P, Bosco G. Middle ear barotrauma during hyperbaric oxygen therapy; a review of occurrences in 5,962 patients. Undersea Hyperb Med. 2019 Mar-Apr-May;46(2):101-106. PMID 31051054